CLINICAL TRIAL: NCT06947382
Title: Multicenter, Case-Control Clinical Validation Study of a Multiplex Blood Protein Biomarker Test, IMMNOV-2, for Early Detection of Pancreatic Ductal Adenocarcinoma (PDAC) in High-Risk Patients
Brief Title: Clinical Validation of Immunovia Next-Generation Blood Biomarker Test to Detect Early-Stage Pancreatic Cancer
Acronym: CLARITI
Status: Completed | Type: Observational
Sponsor: Immunovia, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CLARITI-10
Record Dates: First submitted 2025-04-11; First posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Pancreatic Cancer Stage I; Pancreatic Cancer Stage II; Cancer Diagnosis; PDAC - Pancreatic Ductal Adenocarcinoma
Keywords: PDAC; pancreatic cancer; early detection; Pancreatic Cancer Stage I; Pancreatic Cancer Stage II; pancreatic cancer diagnosis; pancreatic ductal adenocarcinoma; pancreatic cancer detection
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- PDAC Cases: Serum samples from patients recently diagnosed with Stage I or Stage II pancreatic adenocarcinoma (PDAC) with no prior treatment for disease
- Control: Serum samples from non-pancreatic adenocarcinoma (PDAC) patients at high-risk for disease due to familial or genetic history or clinical symptoms.

SUMMARY:
This is a case-control study to clinically validate the performance of a protein biomarker test to differentiate Stage I and Stage II pancreatic ductal adenocarcinoma (PDAC) patient samples from samples acquired from control patients not diagnosed with PDAC but at increased risk of disease due to familial/genetic history or clinical symptoms.

DETAILED DESCRIPTION:
This case-control study is being conducted to determine the performance of a multiplex protein biomarker model in human serum samples.

Serum samples were collected for analysis from patients with Stages I and II pancreatic ductal adenocarcinoma (PDAC) and non-PDAC controls of similar demographics who were at increased risk of PDAC because their familial or genetic history or clinical symptoms. Investigators and patients will not receive individual patient results, therefore patient care will not be impacted by test results.

Analysis of blood samples will be conducted in Immunovia's laboratory in Durham, NC by personnel who are blinded to subject data. Biomarker results will be analyzed using three predefined (locked) algorithm with predefined (locked) cut-offs resulting in a positive/negative test outcome.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent available
* > 45 years of age
* PDAC cases

  * Treatment-naïve, pathologically confirmed PDAC Stage I or Stage II
  * Sporadic or familial/genetic PDAC
* Controls

  * Individuals at high risk for PDAC because of their familial and/or genetic history
  * Individuals with clinical symptoms/signs (e.g. abnormal imaging of the pancreas such as fullness, unexplained weight loss, etc) suggestive of PDAC who were found to NOT have PDAC based on clinical investigation (imaging evidence within 6 months of blood draw)
  * Controls will be selected to have similar demographic features (age/gender) to PDAC patients, as possible.

Exclusion Criteria:

* Prior treatment for PDAC (i.e., prior resection, radiotherapy, or chemotherapy)
* Current immunosuppressive (e.g. systemic steroid therapy) or chemotherapy
* Major surgery or significant trauma within 12 weeks prior to blood sample collection
* Non-PDAC malignancies within 3 years prior to sample collection squamous or basal cell skin carcinoma is not an exclusion criteria)
* Control patients who currently have

  * biliary obstruction secondary to gallstones
  * prior diagnosis or imaging evidence of chronic pancreatitis
  * cystic pancreatic lesions >3.0 cm in diameter or showing worrisome features according to Fukuoka Consensus Guidelines.

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Samples will be retrospectively obtained under the Immunovia PanDetect, PanFam or PRECEDE study protocols, or unique institutional protocols for sample collection through high-risk PDAC surveillance programs.
Sampling Method: Non-Probability Sample
Enrollment: 1066 (Actual)
Dates: Start 2024-09-02 (Actual); Primary Completion 2024-12-09 (Actual); Study Completion 2025-01-06 (Actual)

PRIMARY OUTCOMES:
Determine the sensitivity and specificity of IMMNOV-2 to differentiate serum samples from patients diagnosed with PDAC and controls. | Baseline

SECONDARY OUTCOMES:
Sensitivity and specificity of IMMNOV-2 compared to sensitivity and specificity of CA19-9 alone in the overall population | Baseline
Sensitivity and specificity of IMMNOV-2 in patients age > or equal to 65 years of age | Baseline
Sensitivity and specificity of IMMNOV-2 compared to sensitivity and specificity of CA19-9 alone in patients age > or equal to 65 years old | Baseline

CONTACTS AND LOCATIONS:
Locations (15):
- United States (12):
  - HonorHealth Clinical Research Institute, Scottsdale, Arizona
  - St. John's Cancer Institute, Burbank, California
  - University of California San Diego, La Jolla, California
  - Stanford Gastroenterology and Hepatology, Stanford, California
  - University of Miami, Miami, Florida
  - University of Chicago Medical Center, Chicago, Illinois
  - Mount Sinai Hospital, New York, New York
  - Oregon Health Sciences University, Portland, Oregon
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Regional One Health, Memphis, Tennessee
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
- The Research Institute of the McGill University Health Centre, Montreal, Canada
- University of Verona, Verona, Italy
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No
Individual patient results will not be shared with patients.